CLINICAL TRIAL: NCT06111937
Title: Correlation Between Time Interval After Gastric Emptying With Ultrasound Assessment and Quality of Bowel Cleansing in Patients Undergoing Painless Colonoscopy: a Randomized, Prospective, Controlled Trial
Brief Title: Time Interval After Gastric Emptying and Quality of Bowel Cleansing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KY20230428-01
Record Dates: First submitted 2023-09-21; First posted 2023-11-01 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2024-03

CONDITIONS: Colonoscopy
Keywords: Colonoscopy; Ultrasound

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colonoscopy within 2-4 h (Experimental): Patients received ultrasound gastric assessment every 15 minutes 2 hours immediately after taking the last dose of MgSO4 solution. During this period, if the gastric ultrasound assessment showed that the patient had an "empty stomach", and painless colonoscopy was performed within 2 hours while the gastric is empty.
  Interventions: Other: after ultrasound gastric assessment to ensure gastric empty, painless colonoscopy was performed within 2 hours
- colonoscopy within 4-6 h (No Intervention): The patients received ultrasound gastric assessment every 15min 4h immediately after taking the last dose of MgSO4 solution on the examination day, and colonoscopy was to completed within 4-6h after taking the MgSO4 solution if the gastric ultrasound assessment showed that the patient had an "empty stomach".

INTERVENTIONS:
Other: after ultrasound gastric assessment to ensure gastric empty, painless colonoscopy was performed within 2 hours — Patients received gastric ultrasound examination every 15 minutes 2 or 4 hours immediately after taking the last dose of MgSO4 solution in group A or B respectively.
  Other Names: Ultrasound gastric assessment
  Arms: colonoscopy within 2-4 h

SUMMARY:
The goal of this [clinical trial] is to [explore the balance time point between the waiting time for intestinal preparation after gastric emptying and quality of bowel preparation.] in [patients with painless colonoscopy]. The main question[s] it aims to answer are:

[whether the gastric is empty or not 2 hours after finishing drinking 1.5 L of MgSO4 solution within 2 hours] [whether the quality of patients' bowel preparation is superior in a time period of 2-4 hours after finishing drinking 1.5 L of MgSO4 solution] Participants will [ be asked finishing the last dose of 1.5 L MgSO4 solution within 2 hours and received ultrasound gastric assessment immediately 2 or 4 hours after finishing drinking MgSO4 solution in a 15 minutes time interval until the gastric is empty. As soon as the gastric is empty, patients receive painless colonoscopy within 2 hours or 2-4 hours.

Researchers will compare [patients receiving painless colonoscopy within 2 hours or 2-4 hours after finishing drinking 1.5 L of MgSO4 solution] to see if [the quality of patients' bowel preparation is superior in a time period of within 2 hours].

DETAILED DESCRIPTION:
All subjects ate a light diet the day before the examination and fasted after 19:00 on the night before examination. A segmented intestinal cleansing regimen of 3L MgSO4 was adopted: 1.5L was taken one night before the examination; On the day of the examination, the second dose of 1.5L was taken and finished within 2 hours. The medication method was guided by professional nursing staff. All subjects were instructed to take appropriate activities during the administration of intestinal cleanser to promote excretion. Patients were divided into two groups (group A and group B) using random number table method. Patients in group A received gastric ultrasound examination every 15 minutes 2 hours immediately after taking the last dose of MgSO4 solution. During this period, if the gastric ultrasound showed that the patient had an "empty stomach", and painless colonoscopy was performed within 2 hours while the gastric is empty. If the gastric ultrasound still showed "full stomach" at 4h, the patient was abandoned, but gastric ultrasound assessment continued until the stomach was empty. The patients in group B received gastric ultrasound examination every 15min 4h immediately after taking the last dose of MgSO4 solution on the examination day, and colonoscopy was to completed within 4-6h after taking the MgSO4 solution if the gastric ultrasound showed that the patient had an "empty stomach". If the gastric ultrasound still shows "full stomach" at 6h, it is eliminated, but continuing to perform gastric ultrasound every 15min until the " stomach was empty ". All patients received general anesthesia by the same senior anesthesiologist using propofol 2 mg/kg and remifentanil 0.2 ug/kg. The BIS value of anesthesia depth was controlled in the range of 40-60, and propofol and remifentanil were added as needed. The same chief gastroenterologist performed the colonoscopy and evaluated the quality of intestinal cleaning.

ELIGIBILITY:
Inclusion Criteria:

1.Patients who receiving elective colonoscopy under general anesthesia

Exclusion Criteria:

1. Patients with severe heart and lung diseases who cannot tolerate anesthesia or colonoscopy
2. chronic constipation
3. history of gastric or intestinal surgery
4. diabetes, Parkinson's disease, stroke,

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Boston bowel preparation quality scale | five minutes after finishing colonoscopy examination
  Using Boston bowel preparation quality scale: 3 score, the intestinal cleaning range is more than 90%, no fecal residue, clear vision, or only some clear liquid exists; 2 score, The intestinal cleaning range was 75% to 90%, only a small amount of intestinal residue or fecal water remained, which had no effect on the examination and observation; 1 score,fecal residue or fecal water exists in more intestinal segments, and can continue to enter the lens after rinsing with water; 0 score: There are more fecal residues in the intestinal cavity, and it is impossible to continue the examination. According to the above scoring criteria, the intestinal cleanliness of the left colon, transverse colon and right colon were scored respectively. The total score ≥6 was considered to be good intestinal preparation. The total score < 6 points was considered that the intestinal preparation was poor.
full stomach rate after finishing MgSO4 solution under different waiting time | 2 or 4 hours after finishing taking MgSO4 solution
  recording full stomach rate using gastric ultrasound

SECONDARY OUTCOMES:
The rate of ileum intubation while performing colonoscopy | while performing colonoscopy
  recording rate of ileum intubation
the detection rate of polyp and adenoma while performing colonoscopy | while performing colonoscopy
  recording the detection rate of polyp and adenoma

CONTACTS AND LOCATIONS:
Overall Officials: Gu JianPing, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee J, Kim TO, Seo JW, Choi JH, Heo NY, Park J, Park SH, Yang SY, Moon YS. Shorter waiting times from education to colonoscopy can improve the quality of bowel preparation: A randomized controlled trial. Turk J Gastroenterol. 2018 Jan;29(1):75-81. doi: 10.5152/tjg.2018.17467. PMID 29391311
- [Result] Tooson JD, Gates LK Jr. Bowel preparation before colonoscopy. Choosing the best lavage regimen. Postgrad Med. 1996 Aug;100(2):203-4, 207-12, 214. doi: 10.3810/pgm.1996.08.59. PMID 8700818
- [Result] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784